CLINICAL TRIAL: NCT07237217
Title: Guided Group Telehealth to Deliver Evidence-based Therapeutic Care to Black College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Veronica Tetterton (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor-Investigator, Dr. Veronica Tetterton, Principal Investigator, The Sweet I AM
Organization: The Sweet I AM (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-44; 1R43MD020009-01 (NIH)
Record Dates: First submitted 2025-11-13; First posted 2025-11-19 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Anxiety Depression
Keywords: mental health; college students; asynchronous group therapy
MeSH Terms: conditions — Psychological Well-Being | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Group Therapy (GGT) via TheraGroup (Experimental): Participants in the GGT group will receive the same psychoeducational information and reading resources about the CBT coping skills and encouragement of reflection on homework assignments in a group online chat environment. Participants in GGT will also receive support in the form of direct asynchronous communication with the therapist and asynchronous communication with peers struggling with similar issues.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT) Coping Skills Training
- Individual Teletherapy (IT) (Active Comparator): Participants in the IT group will receive 1 one 1 teletherapy using the 12-week structured modules. The therapist will be providing psychoeducational information and reading resources about the CBT coping skills and encouragement of reflection on homework assignments in session (via video, audio or text therapy).
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT) Coping Skills Training

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) Coping Skills Training — 12 Week CBT Coping Skills Training Modules

SUMMARY:
The goal of this study is to address the mental health crisis among college students by creating a promising solution for group teletherapy, which is equivalent to individual teletherapy in terms of treatment outcomes.The main question it aims to answer is: if participants' outcome measures in TheraGroup are in line with participants' outcome measures in individual therapy. The goal of the current SBIR is to test TheraGroup, the first large scale virtual group platform for evidenced-based mental health therapy. The TheraGroup application addresses the market surge in the demand for care and the shortage of mental health professionals as it represents an economically viable treatment alternative to individual teletherapy.

DETAILED DESCRIPTION:
Mental illness among college students has become a public health crisis. Even before the pandemic, many college campuses lacked the resources to support students' mental health needs. College campus counseling centers have begun to think creatively about how to meet the growing demand for services as the number of available therapists is insufficient to treat the number of students seeking help. TheraGroup is the solution to leverage innovative group technology to provide Guided Group Therapy (GGT) in which students receive evidenced-based Cognitive Behavioral Therapy (CBT) coping skills training to address the high demand for mental health services and bridge the gap in services on college campuses. TheraGroup is the first large scale virtual group real-time platform for evidenced-based mental health therapy. TheraGroup is a HIPAA-compliant, platform-agnostic tool that provides the channel through which GGT will be facilitated to service college students to improve student mental health outcomes. In Aim 1, researchers will develop the TheraGroup platform. Researchers will achieve this by optimizing the existing platform, which is therapy enabled for one-to-one therapy, to enable one-to-many communication in a large group context. In addition, researchers will develop other proprietary features that create an anonymous and interactive group discussion experience. The proof of concept will be demonstrated with high usage across multiple devices. In Aim 2, researchers will implement a feasibility study to assess the impact of GGT via TheraGroup on measures of engagement, user experience, and mental health outcomes in college students. If participants' outcome measures in the GGT group are in line with participants' outcome measures in the IT group, the feasibility study will serve as a precursor to testing the effects of GGT via TheraGroup using a larger scale randomized control trial. Achieving these aims could suggest TheraGroup is a new actionable tool to supplement existing mental health interventions to address the ever-growing need for mental health services college students.

ELIGIBILITY:
Inclusion Criteria:

* Individuals at PVAMU 18 years and older

Exclusion Criteria:

* Individuals younger than 18 years of age will be excluded from the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2024-09-22 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Completion rate | 12 weeks
  Out of the 40 participants in the clinical trial, how many completed a certain percentage of the 12 week intervention
Engagement with Telehealth Therapy (Custom 8-Item Engagement Scale) | Week 4, 8, and 12
  Engagement will be measured using a custom 8-item self-report scale. Each item is rated from 1 to 5, producing a total score range of 8 to 40. Higher scores indicate better engagement, except for negatively worded items which will be reverse-scored prior to computing the total score. Items assess interest, focus, enjoyment, motivation, clarity, frustration, and perceived boredom.
User Experience Qualitative Feedback (No Numeric Outcome) | Week 4, 8, and 12
  User experience will be assessed through three open-ended qualitative questions evaluating what participants enjoyed, what could be improved, and whether the psychoeducational content felt culturally relevant. These questions do not produce a numeric score.
  User Feedback Experience
  1. What, if anything, did you enjoy about your experience in using the guided telehealth therapy?
  2. What, if anything, could be improved about your experience in using the guided telehealth therapy?
  3. Did you feel the content was culturally relevant to you? Please explain

SECONDARY OUTCOMES:
Generalized Anxiety Disorder-7 (GAD-7) Score | Baseline, Week 4, 8, and 12
  Anxiety symptoms will be assessed using the Generalized Anxiety Disorder 7-Item scale (GAD-7), a self-report measure with 7 items scored from 0 to 3, yielding a total score range of 0 to 21. Higher scores indicate worse anxiety symptoms. The measure assesses nervousness, uncontrollable worry, overthinking, restlessness, irritability, difficulty relaxing, and fear of impending harm.
Patient Health Questionnaire -9 (PHQ-9) Score | Baseline, Week 4, 8, and 12
  Depression symptoms will be assessed using the Patient Health Questionnaire 9-Item (PHQ- 9), a self-report scale with 9 items scored from 0 to 3, yielding a total score range of 0 to 27. Higher scores indicate worse depressive symptoms. The measure assesses anhedonia, low mood, sleep disturbance, fatigue, appetite changes, self-worth, concentration, psychomotor changes, and suicidal thoughts.

CONTACTS AND LOCATIONS:
Locations (1):
- PVAMU, Prairie View, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
For confidentiality purposes.

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2025-01-31): https://cdn.clinicaltrials.gov/large-docs/17/NCT07237217/Prot_ICF_002.pdf
  • Statistical Analysis Plan (2025-03-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT07237217/SAP_003.pdf